CLINICAL TRIAL: NCT00005813
Title: A Phase I Trial of Intratumoral Bispecific Antibody and Activated Monocytes in Patients With Recurrent or Refractory Glioblastoma Multiforme
Brief Title: Bispecific Antibody Plus White Blood Cells in Treating Patients With Recurrent or Refractory Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: D9705; P30CA023108 (NIH); NCI-G00-1783 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2000-06-02; First posted 2003-05-20 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bispecific antibody MDX447
Biological: lymphokine-activated killer cells
Procedure: conventional surgery

SUMMARY:
RATIONALE: Bispecific antibodies plus white blood cells may be able to locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of combining bispecific antibodies with white blood cells in treating patients who have recurrent or refractory glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the safety and tolerability of bispecific antibody MDX447 and activated monocytes in patients with recurrent or refractory glioblastoma multiforme.
* Determine the response, time to tumor progression, and overall survival of these patients treated with this regimen.

OUTLINE: This is a dose escalation study.

Patients undergo maximal surgical debulking of the tumor at the time of reservoir placement. Within 2-4 weeks after surgery, patients receive one treatment of intratumoral bispecific antibody MDX447 and activated monocytes. Stable or responding patients may receive a second treatment 1 month later.

Cohorts of 1 or 3 patients receive escalating doses of bispecific antibody MDX447 and activated monocytes until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: A total of 13 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven glioblastoma multiforme with evidence of epidermal growth factor receptor (EGFR) expression on tumor cell surfaces

  * No astrocytoma, anaplastic astrocytoma, or oligodendroglioma
  * No infratentorial or multifocal tumor
* Recurrence or progression following at least one prior therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Greater than 2 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* ALT, AST, and alkaline phosphatase no greater than 2.5 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 2.0 times ULN

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other medical or psychiatric illness that would preclude study
* No other concurrent malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas)

Endocrine therapy:

* Concurrent steroid therapy allowed

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-03; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilo E Fadul, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States